CLINICAL TRIAL: NCT01698320
Title: A Multi-Center 52-Week Study to Assess the Safety of Albuterol Spiromax® in Subjects With Asthma
Brief Title: Safety Study of Albuterol Spiromax® in Subjects With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABS-AS-307
Record Dates: First submitted 2012-09-14; First posted 2012-10-03 (Estimated); Results first posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo MDPI-Albuterol MDPI (Placebo Comparator): During the 12-week double-blind period, participants take 2 inhalations of placebo MDPI (multi-dose dry powder inhaler), four times a day (QID) at approximately 7:00 AM, 12:00 PM, 5:00 PM, and bedtime.
  The double-blind period is followed by a 40-week open-label period in which all study participants take albuterol MDPI 90 micrograms/inhalation, 2 inhalations every 4-6 hours as needed (PRN) and, if applicable, 2 inhalations 15-30 minutes prior to sports/exercise.
  Interventions: Drug: Placebo MDPI; Drug: Albuterol MDPI
- Albuterol MDPI-Albuterol MDPI (Experimental): During the 12-week double-blind period, participants take 2 inhalations of albuterol MDPI (multi-dose dry powder inhaler or Spiromax®) 90 mcg/inhalation, four times a day (QID) at approximately 7:00 AM, 12:00 PM, 5:00 PM, and bedtime for a total daily dose of 720 micrograms per day.
  The double-blind period is followed by a 40-week open-label period in which all study participants take albuterol MDPI 90 micrograms/inhalation, 2 inhalations every 4-6 hours as needed (PRN) and, if applicable, 2 inhalations 15-30 minutes prior to sports/exercise.
  Interventions: Drug: Albuterol MDPI

INTERVENTIONS:
Drug: Placebo MDPI — Placebo MDPI (multi-dose dry powder inhaler) to match the active intervention.
  Other Names: placebo
  Arms: Placebo MDPI-Albuterol MDPI
Drug: Albuterol MDPI — Albuterol MDPI (multi-dose dry powder inhaler or Spiromax®) 90 mcg/inhalation.
  Other Names: ProAir® RespiClick; Albuterol Spiromax

SUMMARY:
The purpose of this study is to evaluate the safety of Albuterol Spiromax® over 52 weeks during two dosing periods: (1) a 12-week, double-blind, placebo-controlled QID dosing period followed by (2) a 40-week, open-label PRN dosing period, and to evaluate Albuterol Spiromax® device performance through the life of the device during the study.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA signed and dated by the subject or written informed assent signed and dated both by the subject and/or parent/caregiver/legal guardian before conducting any study related procedure.
* Males or females with asthma ages 12 years or older at screening.
* Documented history of persistent asthma and current use of an MDI containing any short-acting beta-adrenergic agonist (e.g. albuterol, levalbuterol,) on average of at least once/week over the 4-weeks prior to screening. The asthma diagnosis must be consistent with the diagnosis of asthma as per the National Asthma Education and Prevention Program.
* If female, is currently not pregnant, breast feeding, or attempting to become pregnant (for 4 weeks before the screening visit and throughout the duration of the study), and is of Non-childbearing potential, defined as:

  * ≥1 year post-menopausal or
  * Surgically sterile (tubal ligation, bilateral oophorectomy, salpingectomy, or hysterectomy) or is of
  * Childbearing potential, has a negative serum pregnancy test, and is willing to commit to using a consistent and acceptable method of birth control
* General good health in the opinion of the investigator as indicated by medical history, physical examination, laboratory tests (hematology, serum chemistry and urinalysis) assessed as either normal or abnormal not clinically significant (NCS) per the principal investigator, as well as a 12-lead ECG interpreted as either "Normal" or "Abnormal NCS" as determined by the central cardiologist. Subjects must also be free of any clinically significant, uncontrolled concomitant conditions other than asthma that could interfere with study conduct, influence the interpretation of study observations/results, or put the subject at increased risk during the trial.
* Capable of understanding the requirements, risks, and benefits of study participation, and, as judged by the investigator, and being compliant with all study requirements (visits, record-keeping, etc).
* Non-smoker for at least one year prior to the screening visit and a maximum pack-year (PY) smoking history of 10 years.
* Able to demonstrate proper inhaler technique with study inhaler.

Exclusion Criteria:

* Pregnancy, nursing, or plans to become pregnant or donate gametes (ova or sperm) for in vitro fertilization during the study period or for 30 days following the subject's last study related visit.
* Participation in any investigational drug trial within 30 days preceding the screening visit or planned participation in another investigational drug trial at any time during this trial.
* A known hypersensitivity to albuterol or any of the excipients in the formulations.
* History of severe milk protein allergy
* History of an upper or lower respiratory tract infection or disorder (including, but not limited to bronchitis, pneumonia, acute or chronic sinusitis, otitis media, influenza, etc) which is not resolved at least 1 week prior to the SV.
* History of alcohol or drug abuse within two years preceding the SV.
* Use of any protocol prohibited concomitant medications for asthma (any oral β2-adrenergic agonists) or any protocol prohibited concomitant non-asthma medications including treatment with β2-adrenergic receptor antagonists and non-selective β-receptor blocking agents such as β-blocking anti-hypertensive products (administered by any route), MAO inhibitors, and/or tricyclic antidepressants. (Subject's own MDI short-acting β-agonist rescue inhaler should be used until the start of the Run-In period when a study rescue inhaler is provided.)
* Inability or unwillingness to comply with the protocol requirements.
* History of life-threatening asthma [defined here as an asthma episode requiring intubation and/or associated with hypercapnea, respiratory arrest or hypoxic seizures.]
* Any asthma exacerbation within 3 months of the SV requiring oral or systemic corticosteroids or any hospitalization for asthma within 6 months of the SV.

Note: An exacerbation of asthma is defined as any worsening of asthma requiring any treatment other than rescue albuterol or the subject's regular asthma maintenance therapy. This includes requiring the use of systemic corticosteroids and/or emergency room visit or hospitalization or a change in subject's regular asthma maintenance treatment. A subject does not need to be withdrawn from the study due to an asthma exacerbation unless hospitalization is required or unless the principal investigator believes it is in the subjects' best interest to withdraw from the study.

* Previous participation in an inhaled Albuterol Spiromax® (Teva) study, with the exception of the ABS-AS-306 study.
* Study participation by clinical investigator site employees and/or their immediate relatives.
* Study participation by related or non-related individuals living in the same household, i.e. only one subject per household may participate in the study.
* Any clinically significant endocrine, hematological, hepatic, renal, gastrointestinal, neurological, cardiac, metabolic, immunological, any non-asthmatic acute or chronic pulmonary condition (including but not limited to bronchitis, emphysema, active tuberculosis, bronchiectasis, cystic fibrosis), and malignancy other than basal cell carcinoma. Significant is defined for this protocol as any condition that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which could affect the safety analyses.
* Any medical or psychological condition that in the investigator's opinion should preclude enrollment.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - Teva Investigational Site 10169, Huntington Beach, California
  - Teva Investigational Site 10157, San Diego, California
  - Teva Investigational Site 10148, Denver, Colorado
  - Teva Investigational Site 10159, Denver, Colorado
  - Teva Investigational Site 10158, Miami, Florida
  - Teva Investigational Site 10168, Miami, Florida
  - Teva Investigational Site 10154, Gainesville, Georgia
  - Teva Investigational Site 10161, Louisville, Kentucky
  - Teva Investigational Site 10162, Bethesda, Maryland
  - Teva Investigational Site 10166, Wheaton, Maryland
  - Teva Investigational Site 10151, Minneapolis, Minnesota
  - Teva Investigational Site 10142, Plymouth, Minnesota
  - Teva Investigational Site 10152, St Louis, Missouri
  - Teva Investigational Site 10146, Bellevue, Nebraska
  - Teva Investigational Site 10160, Skillman, New Jersey
  - Teva Investigational Site 10144, Rochester, New York
  - Teva Investigational Site 10141, High Point, North Carolina
  - Teva Investigational Site 10153, Raleigh, North Carolina
  - Teva Investigational Site 10147, Canton, Ohio
  - Teva Investigational Site 10143, Cincinnati, Ohio
  - Teva Investigational Site 10167, Sylvania, Ohio
  - Teva Investigational Site 10150, Eugene, Oregon
  - Teva Investigational Site 10156, Portland, Oregon
  - Teva Investigational Site 10155, El Paso, Texas
  - Teva Investigational Site 10149, New Braunfels, Texas
  - Teva Investigational Site 10145, San Antonio, Texas
  - Teva Investigational Site 10170, San Antonio, Texas
  - Teva Investigational Site 10163, Burke, Virginia
  - Teva Investigational Site 10165, Seattle, Washington
  - Teva Investigational Site 10164, Greenfield, Wisconsin

REFERENCES:
- [Derived] Raphael G, Taveras H, Iverson H, O'Brien C, Miller D. Twelve- and 52-week safety of albuterol multidose dry powder inhaler in patients with persistent asthma. J Asthma. 2016;53(2):187-93. doi: 10.3109/02770903.2015.1070862. Epub 2015 Sep 15. PMID 26369589

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 33 patients who were screened but not enrolled, 28 were excluded on the basis of inclusion/exclusion criteria, 2 patients withdrew consent, and 3 patients were lost to follow-up before the baseline visit.
Groups:
- All Enrolled Subjects: Includes subjects who were enrolled in study and participated in the single-blind (subjects were blinded) run-in period in which subjects used the inhaler with placebo and maintained the diary for about one week prior to randomization and starting the 12-week double-blind period.
Period: Run-In Period (Week -1 to Day 0)
Arm/Group | All Enrolled Subjects | Placebo MDPI-Albuterol MDPI | Albuterol MDPI-Albuterol MDPI
Started | 364 | 0 | 0
Completed | 337 | 0 | 0
Not Completed | 27 | 0 | 0
Not completed — Inclusion/exclusion criteria | 24 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Other | 1 | 0 | 0
Period: 12-Week Double-Blind Period
Arm/Group | All Enrolled Subjects | Placebo MDPI-Albuterol MDPI | Albuterol MDPI-Albuterol MDPI
Started | 0 | 169 | 168
Safety Population | 0 | 170 (One participant took both placebo and albuterol so is counted in both treatment groups for safety.) | 168
Completed | 0 | 165 | 156
Not Completed | 0 | 4 | 12
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 2
Not completed — Protocol Violation | 0 | 0 | 2
Not completed — Pregnancy | 0 | 1 | 1
Not completed — Sponsor requested subject withdrawal | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 4
Period: 40-Week Open-Label Period
Arm/Group | All Enrolled Subjects | Placebo MDPI-Albuterol MDPI | Albuterol MDPI-Albuterol MDPI
Started | 0 | 165 | 156
Completed | 0 | 146 | 146
Not Completed | 0 | 19 | 10
Not completed — Adverse Event | 0 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 11 | 7
Not completed — Pregnancy | 0 | 2 | 1
Not completed — Sponsor requested subject withdrawal | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set of randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo MDPI-Albuterol MDPI | Albuterol MDPI-Albuterol MDPI | Total
Number analyzed (Participants) | 169 | 168 | 337
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (15.14) | 36.6 (15.04) | 36.8 (15.07)
Age, Customized [Number; unit: participants]
  12-17 years | 19 | 25 | 44
  18-64 years | 143 | 135 | 278
  65+ years | 7 | 8 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 103 | 214
  Male | 58 | 65 | 123
Race/Ethnicity, Customized [Number; unit: participants]
  White | 129 | 125 | 254
  Black | 35 | 38 | 73
  Asian | 2 | 4 | 6
  American Indian or Alaskan Native | 2 | 1 | 3
  Pacific Islander | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 25 | 28 | 53
  Not Hispanic or Latino | 144 | 140 | 284
Weight [Mean (Standard Deviation); unit: kg] | 82.3 (21.09) | 81.2 (21.4) | 81.8 (21.22)
Height [Mean (Standard Deviation); unit: cm] | 167.4 (8.67) | 168.6 (9.52) | 168.0 (9.11)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.2 (6.96) | 28.5 (6.81) | 28.8 (6.88)

OUTCOME MEASURES:

1. Primary Outcome: Participants With Adverse Experiences During Weeks 0-12 (Double-Blind Period)
Description: Adverse events (AEs) summarized in this table are those that began or worsened after treatment with study drug (treatment-emergent AEs). An adverse event was defined in the protocol as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= an AE which prevents normal daily activities. Relation of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: Day 1 to Week 12
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Placebo MDPI-Albuterol MDPI | Albuterol MDPI-Albuterol MDPI
Number analyzed (Participants) | 170 | 168
participants
  Any adverse event | 105 | 84
  Severe adverse event | 6 | 3
  Treatment-related adverse event | 1 | 5
  Deaths | 0 | 0
  Other serious adverse events | 1 | 0
  Withdrawn from treatment due to adverse events | 1 | 1

2. Other Pre Specified Outcome: Composite Measurement of Device Ruggedness From Baseline to Week 52
Description: Device Ruggedness: Reports of any problems/malfunction of the device (e.g., lack of efficacy, problems/malfunction after the device is dropped or sustains physical impact).
Time Frame: Baseline to Week 52
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Device Invitro Evaluations to Week 52
Description: Device In Vitro Evaluations - All used study inhalers will be collected and a random selection of inhalers will be tested as follows:
  * Fifty (50) Albuterol Spiromax® inhalers used during weeks 0-12 will be randomly selected for in vitro testing
  * Fifty (50) Albuterol Spiromax® inhalers used during weeks 12-52 will be randomly selected for in vitro performance testing
Time Frame: Baseline to Week 52
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Daily AM Peak Expiratory Flow (PEF) to Week 52
Description: Daily AM PEF will be recorded throughout the duration of the study to provide information on the subject's asthma status in order to assist in distinguishing between the use of back-up rescue medication related to an increased need for asthma symptom relief from that related to an issue with the Albuterol Spiromax® rescue inhaler.
Time Frame: Baseline to Week 52
Reporting Status: Not Posted

5. Primary Outcome: Participants With Adverse Experiences During Weeks 13-52 (Open-Label Period)
Description: as for outcome 1
Time Frame: Weeks 13-52
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Placebo MDPI-Albuterol MDPI | Albuterol MDPI-Albuterol MDPI
Number analyzed (Participants) | 165 | 156
participants
  Any adverse event | 106 | 94
  Severe adverse event | 12 | 13
  Treatment-related adverse event | 2 | 1
  Deaths | 0 | 0
  Other serious adverse events | 3 | 4
  Withdrawn from treatment due to adverse events | 2 | 2

6. Primary Outcome: Electrocardiogram (ECG) Results At Weeks 0, 12, and 52
Description: A standard 12-lead ECG was performed at screening, week 12, and week 52 or early termination/discontinuation. The ECG recording methods were centralized and standardized across all study participants. A centralized cardiologist was responsible for providing all ECG interpretations.
Time Frame: Weeks 0 (screening visit), 12, and 52
Population: Safety population. Participants with assessments at each time point are reported.
Measure: Number; unit: participants
Arm/Group | Placebo MDPI-Albuterol MDPI | Albuterol MDPI-Albuterol MDPI
Number analyzed (Participants) | 170 | 168
participants
  Week 0: Normal | 151 | 154
  Week 0: Abnormal, not clinically relevant | 19 | 14
  Week 0: Abnormal, clinically relevant | 0 | 0
  Week 12: Normal (n=166, 155) | 143 | 140
  Week 12: Abnormal, not clinically relevant | 23 | 15
  Week 12: Abnormal, clinically relevant | 0 | 0
  Week 52: Normal (n=152, 161) | 138 | 148
  Week 52: Abnormal, not clinically relevant | 23 | 13
  Week 52: Abnormal, clinically relevant | 1 | 0

7. Primary Outcome: Change From Baseline in Blood Pressure Measurements to Week 12 and Week 52
Description: Participants were seated at least 2 minutes before blood pressure measurements were obtained by either an electronic or manual sphygmomanometer.
  Week 12 values represent change from Week 0. Week 52 values represent change from Week 12.
Time Frame: Week 0, Week 12 and Week 52
Population: Safety population. Participants with assessments at each time point are reported.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo MDPI-Albuterol MDPI | Albuterol MDPI-Albuterol MDPI
Number analyzed (Participants) | 170 | 168
mmHg
  Systolic BP Week 12 (n=166, 155) | 1.0 (11.27) | 0.2 (10.99)
  Systolic BP Week 52 (n=159, 155) | -0.4 (11.54) | 0.7 (10.31)
  Diastolic BP Week 12 (n=166, 155) | 0.0 (9.16) | 0.3 (7.62)
  Diastolic BP Week 52 (n=159, 155) | 0.2 (9.14) | 1.0 (8.15)

8. Primary Outcome: Change From Baseline in Pulse Measurements to Week 12 and Week 52
Description: Participants were seated at least 2 minutes before pulse measurements were obtained by radial pulse.
  Week 12 values represent change from Week 0. Week 52 values represent change from Week 12.
Time Frame: Week 0, Week 12 and Week 52
Population: Safety population. Participants with assessments at each time point are reported.
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Placebo MDPI-Albuterol MDPI | Albuterol MDPI-Albuterol MDPI
Number analyzed (Participants) | 170 | 168
beats/minute
  Pulse Week 12 (n=166, 155) | -0.1 (9.40) | 0.9 (9.53)
  Pulse Week 52 (n=159, 155) | -0.4 (10.08) | -0.3 (9.77)

9. Primary Outcome: Participants With Abnormal and Clinically Relevant Physical Exam Findings at Weeks 0, 12 and 52
Description: The physical exam was performed by a qualified healthcare professional, and when possible, the same qualified healthcare professional that performed the physical examination at study screening performed all the scheduled physical examinations. Abnormalities and clinical relevance were determined by the qualified healthcare professional.
  HEENT = head, eyes, ears, nose, throat
Time Frame: Weeks 0, 12 and 52
Population: Safety population. Participants with assessments at each time point are reported.
Measure: Number; unit: participants
Arm/Group | Placebo MDPI-Albuterol MDPI | Albuterol MDPI-Albuterol MDPI
Number analyzed (Participants) | 170 | 168
participants
  General appearance - Week 0 (n=170, 167) | 0 | 0
  General appearance - Week 12 (n=166, 155) | 1 | 0
  General appearance - Week 52 (n=162, 161) | 0 | 0
  HEENT - Week 0 (n=170, 167) | 0 | 0
  HEENT - Week 12 (n=166, 155) | 1 | 1
  HEENT - Week 52 (n=162, 161) | 2 | 2
  Chest and lungs - Week 0 (n=170, 167) | 0 | 0
  Chest and lungs - Week 12 (n=166, 155) | 1 | 1
  Chest and lungs - Week 52 (n=162, 161) | 3 | 2
  Heart - Week 0 (n=170, 167) | 0 | 0
  Heart - Week 12 (n=166, 155) | 0 | 0
  Heart - Week 52 (n=162, 161) | 0 | 0
  Abdomen - Week 0 (n=168, 167) | 0 | 0
  Abdomen - Week 12 (n=166, 155) | 0 | 0
  Abdomen - Week 52 (n=162, 161) | 0 | 1
  Musculoskeletal - Week 0 (n=169, 167) | 0 | 0
  Musculoskeletal - Week 12 (n=166, 155) | 0 | 0
  Musculoskeletal - Week 52 (n=162, 161) | 0 | 0
  Skin - Week 0 (n=169, 167) | 0 | 0
  Skin - Week 12 (n=167, 155) | 0 | 0
  Skin - Week 52 (n=162, 161) | 0 | 0
  Lymph Nodes - Week 0 (n=169, 167) | 0 | 0
  Lymph Nodes - Week 120 (n=166, 155) | 0 | 0
  Lymph Nodes - Week 52 (n=162, 161) | 0 | 0
  Neurological - Week 0 (n=169, 167) | 0 | 0
  Neurological - Week 12 (n=166, 155) | 0 | 0
  Neurological - Week 52 (n=162, 161) | 0 | 0
  Extremities/back - Week 0 (n=169, 167) | 0 | 0
  Extremities/back - Week 12 (n=166, 155) | 0 | 0
  Extremities/back - Week 52 (n=162, 160) | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Week 52
Groups:
- Albuterol MDPI - Double-blind Period: Albuterol multi-dose dry powder inhaler (MDPI or Spiromax) at a dose of 720 micrograms per day administered as 2 inhalations of 90 mcg /inhalation four times a day for the 12 week double-blind period.
- Placebo MDPI - Double-blind Period: Placebo delivered using a multi-dose dry powder inhaler (MDPI or Spiromax) as 2 inhalations four times a day for the 12 week double-blind period.
- Albuterol MDPI (Formerly Placebo) - Open Label Period: After completing 12 weeks of placebo QID treatment, participants continue into the 40 week open-label period in which they administer albuterol multi-dose dry powder inhaler (Spiromax) inhalations of 90 mcg/inhalation as required (PRN).
- Albuterol MDPI (Formerly Albuterol) - Open Label Period: After completing 12 weeks of albuterol QID treatment, participants continue into the 40 week open-label period in which they administer albuterol multi-dose dry powder inhaler (Spiromax) inhalations of 90 mcg/inhalation as required (PRN).
Arm/Group | Albuterol MDPI - Double-blind Period | Placebo MDPI - Double-blind Period | Albuterol MDPI (Formerly Placebo) - Open Label Period | Albuterol MDPI (Formerly Albuterol) - Open Label Period
Serious Adverse Events (participants affected / at risk) | 0/168 | 1/170 | 3/169 | 4/168
Other Adverse Events (participants affected / at risk) | 51/168 | 80/170 | 64/169 | 67/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albuterol MDPI - Double-blind Period (N=168) | Placebo MDPI - Double-blind Period (N=170) | Albuterol MDPI (Formerly Placebo) - Open Label Period (N=169) | Albuterol MDPI (Formerly Albuterol) - Open Label Period (N=168)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albuterol MDPI - Double-blind Period (N=168) | Placebo MDPI - Double-blind Period (N=170) | Albuterol MDPI (Formerly Placebo) - Open Label Period (N=169) | Albuterol MDPI (Formerly Albuterol) - Open Label Period (N=168)
Bronchitis (Infections and infestations) | 3 (4) | 9 (10) | 6 (7) | 6 (6)
Influenza (Infections and infestations) | 3 (3) | 10 (11) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 10 (12) | 17 (22) | 16 (20) | 20 (26)
Sinusitis (Infections and infestations) | 8 (9) | 13 (14) | 10 (11) | 19 (23)
Upper respiratory tract infection (Infections and infestations) | 23 (26) | 31 (36) | 27 (36) | 15 (16)
Headache (Nervous system disorders) | 10 (19) | 12 (16) | 8 (25) | 10 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 12 (13) | 18 (19) | 11 (14)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 11 (11) | 10 (12) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.